CLINICAL TRIAL: NCT06816927
Title: A Multi-Center, Randomized, Phase 2 Trial of Glioblastoma Immunotherapy Advancement With Nivolumab and Relatlimab (GIANT)
Brief Title: Trial of Glioblastoma Immunotherapy Advancement With Nivolumab and Relatlimab
Acronym: GIANT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Principal Investigator, Mustafa Khasraw, MBChB, MD, FRCP, FRACP, Professor of Neurosurgery • Neuro Oncology, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00116940
Record Dates: First submitted 2024-12-18; First posted 2025-02-10 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Newly Diagnosed Glioblastoma
MeSH Terms: interventions — Nivolumab; relatlimab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab (Experimental): 4 stages of treatment on Arm 1 are:
  1. Neoadjuvant Treatment: Patient will receive a single dose of 480 mg by IV infusion on Day 1.
  2. Resection
  3. Part 1 Adjuvant Treatment: Patient will receive 480 mg of nivolumab and 380 mg of relatimab for up to 12 cycles with concomitant radiation 2Gy/day (60 Gy in total). All MGMT methylated patients under Part 1 Adjuvant Treatment setting will also receive 75 mg/m2 TMZ from Day 1 to Day 42 orally.
  4. Part 2 Adjuvant Treatment: Part 1 Adjuvant Treatment will continue without concomitant radiation.
  Interventions: Drug: Nivolumab; Drug: TMZ; Radiation: Radiation Therapy
- Nivolumab and Relatlimab (Experimental): In Arm 2 and Safety Lead-In phase, patients will receive treatment in 4 stages as below:
  1. Neoadjuvant Treatment: Patient will receive a single dose of 480 mg by IV infusion with 480 mg of relatimab on Day 1.
  2. Resection
  3. Part 1 Adjuvant Treatment: Patient will receive 480 mg of nivolumab and 480 mg of relatimab for up to 12 cycles with concomitant radiation 2Gy/day (60 Gy in total). All MGMT methylated patients under Part 1 Adjuvant Treatment setting will also receive 75 mg/m2 TMZ from Day 1 to Day 42 orally.
  4. Part 2 Adjuvant Treatment: Part 1 Adjuvant Treatment will continue without concomitant radiation.
  Interventions: Drug: Nivolumab; Drug: Relatlimab; Drug: TMZ; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Nivolumab — For Neoadjuvant treatment, on both Arms 1 and 2, all 92 patients will receive single dose of 480 mg by IV infusion on Day 1 followed by surgery. Post-resection, in Part 1 Adjuvant treatment, all patients will receive two doses of 480 mg of nivolumab by IV infusion on Days 1 and 29. In Part 2 Adjuvant Treatment of Nivolumab dosing will continue for up to 12 cycles. Each cycle is 28 Days long.
Drug: Relatlimab — For Neoadjuvant treatment, only on Arm 2, 69 patients will receive a single dose of 480 mg of nivolumab and 480 mg of relatimab by IV infusions on Day 1 followed by surgery. Post resection in Part 1 Adjuvant treatment, all patients will receive two doses of 480 mg of nivolumab and relatlimab by IV infusion on Days 1 and 29. In Part 2 Adjuvant Treatment of Relatimab dosing will continue for up to 12 cycles. Each cycle is 28 Days long.
  Arms: Nivolumab and Relatlimab
Drug: TMZ — All patients in safety lead-in, Arm 1 and Arm 2 post resection in Part 1 Adjuvant Treatment setting will receive 75 mg/m2 TMZ from Day 1 to Day 42 orally. In Part 2 Adjuvant Treatment of TMZ dosing with TMZ will continue for up to 6 cycles with 150 mg/m2 for cycle 3 and escalating to 200 mg/m2 for cycles 4 to 8 day 1 to 5 for these 6 cycles.
Radiation: Radiation Therapy — All patients in safety lead-in, Arm 1 and Arm 2 post resection in Part 1 Adjuvant Treatment will receive External Beam Radiation 2 Gy/day (60 Gy in total) Once daily, 5 days per week, for 6 weeks Starting on Day 1

SUMMARY:
GIANT is an open-label, multi-center, randomized, perioperative (neoadjuvant followed by adjuvant), phase 2 trial with a safety lead-in phase to investigate the feasibility, safety and tolerability, and establish the biological activity of nivolumab with or without relatlimab in patients with isocitrate dehydrogenase (IDH) wildtype newly diagnosed glioblastoma (ndGBM).

DETAILED DESCRIPTION:
Hypotheses for GIANT: A perioperative trial of nivolumab with or without relatlimab in patients with ndGBM is feasible and safe and that we will be able to evaluate the biological effect (pharmacodynamics [PD]) of nivolumab monotherapy and in combination with relatlimab in this setting and determine whether there is sufficient biological activity in patients with GBM to warrant further development.

Patients with a ndGBM and those with a previous diagnosis of GBM who have not received prior radiation (RT) or systemic therapy will have histological confirmation of diagnosis either by on study stereotactic biopsy or from an archival tissue. Cohorts of 6 patients will be accrued to receive nivolumab and relatlimab combined with RT and TMZ in the safety lead-in portion. Once determined safe, the randomized portion of the study will commence and patients will be randomized to one of two arms for neoadjuvant treatment prior to surgical resection of their tumor using an unbalanced 1:3 treatment allocation: Arm 1 - nivolumab alone or Arm 2 - nivolumab and relatlimab (combination formulation). After tumor resection, all patients will undergo Part 1 adjuvant treatment and receive RT and temozolomide (TMZ) (TMZ will be omitted in MGMT unmethylated patients), in combination with nivolumab and relatlimab. Afterwards, patients will undergo Part 2 adjuvant treatment, wherein they will receive TMZ in combination with nivolumab and relatlimab until progression or discontinuation criteria are met. All patients will be followed for 2 years after the last patients has been registered.

Primary Objectives:

1. Stage 1 - Safety Lead-In: To assess the safety of concurrently administering nivolumab, relatlimab, RT, with or without TMZ during Part 1 of the Adjuvant Treatment phase in ndGBM patients, with a specific go-no go focus on MGMT methylated patients receiving TMZ
2. Stage 2 - Randomized Phase 2: To assess the feasibility of undertaking a peri-operative study involving administration of nivolumab with or without relatlimab in patients with ndGBM
3. To establish the biological activity of nivolumab administered with or without relatlimab in patients with ndGBM, by demonstrating the presence of tumor infiltrating lymphocytes (TILs) in the resected tumor

Secondary Objectives:

1. To describe the toxicity of nivolumab administered with or without relatlimab during the neoadjuvant phase in patients with ndGBM following tumor biopsy, and prior to surgical resection of their tumor
2. To assess the safety of planned craniotomy and tumor resection performed after biopsy and neoadjuvant treatment with nivolumab administered with or without relatlimab in patients with ndGBM
3. To determine the toxicity of nivolumab administered with relatlimab during the adjuvant phase, following surgical resection of their tumor in patients with ndGBM To assess the pharmacokinetics (PK) of nivolumab administered with or without relatlimab during the neoadjuvant phase following biopsy, and prior to tumor resection for patients with ndGBM
4. To estimate the radiological response rate of nivolumab administered with or without relatlimab in ndGBM
5. To describe survival of patients who have been assigned (as in the Stage 1 safety lead-in) or randomized (Stage 2) to receive neoadjuvant nivolumab administered with or without relatlimab.

After their biopsy or confirmation of diagnosis from the archival tissue, patients will be randomized in the Neoadjuvant Treatment stage to receive one cycle of either nivolumab alone (Arm 1) or the combination of nivolumab and relatlimab (Arm 2). Within 14 (±3) days of day 1 of neoadjuvant treatment all patients registered in Stages 1 and 2 will undergo tumor resection and placement of Ommaya reservoir. After surgery, patients will enter the Part 1 Adjuvant Treatment phase and will receive RT and TMZ chemotherapy in combination with nivolumab and relatlimab. After the last dose of treatment in Part 1 Adjuvant Treatment, patients will begin the Part 2 Adjuvant Treatment phase and will receive 6 cycles of TMZ in combination with nivolumab and relatlimab. Patients that complete the treatment (i.e., complete 12 cycles of nivolumab and relatlimab with or without TMZ in the Part 2 Adjuvant Treatment Phase) or that discontinue treatment for any reason will have an End of Treatment visit and a Safety Follow-up visit 135 days after the End of Treatment visit

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent approved by the IRB
2. Adults ≥ 18 years of age
3. Patients with either:

   * A newly suspected diagnosis of GBM based on MRI
   * A previous diagnosis of GBM and who have not received prior RT or systemic therapy for their brain tumor
4. Patients who in the opinion of the treating neurosurgeon require resection
5. Patient is willing to undergo planned surgical procedures
6. Patient agrees to make biospecimens that will be prospectively collected (after date of consent) available for research
7. Patients who have undergone a diagnostic biopsy or open surgical procedure prior to enrolling in this study:

   * If adequate archival tissue, defined as at least 3 blocks, is readily available, there is clear documentation of its availability, and the patient must consents to provide that tissue, the patient does not need to undergo another biopsy prior to, or on study, in order to be eligible for this trial
   * If archival tissue is sufficient as described above, patient must have either residual enhancing disease requiring resection, or molecularly confirmed GBM with a clear clinical indication for additional resection, as determined by the country PI (or delegate) and the designated trial surgeon.
   * If archival tissue is insufficient, or if the patient previously underwent a needle biopsy and there is no clear documentation of tissue availability, and the patient wishes to enroll, the patient must agree to undergo a repeat biopsy as part of this study prior to Screening.
8. Hematological function as follows:

   * Absolute neutrophil count ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Haemoglobin > 90 g/L
   * Prothrombin time (PT) or partial thromboplastin time (PTT) < 1.5 x upper limit of normal (ULN)
9. Renal function as follows:

   • Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 40 ml/min using the Cockcroft-Gault formula (Appendix 1)
10. Hepatic function as follows:

    * Total bilirubin ≤ 1.5 x ULN (Exception: Patient has known or suspected Gilbert's Syndrome for which additional lab testing of direct and/or indirect bilirubin supports this diagnosis. In these instances, a total bilirubin of ≤ 3.0 x ULN is acceptable)
    * Alkaline phosphatase (ALP) ≤ 2.5 x ULN
    * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
    * Serum albumin ≥ 25 g/L
11. Eastern Co-operative Oncology Group (ECOG) performance status of 0-1 (Appendix 2)
12. Life expectancy of at least 12 months
13. Negative human immunodeficiency virus (HIV) test at Screening
14. Negative hepatitis B surface antigen (HbsAg) test at Screening or positive test followed by a negative hepatitis B virus (HBV) DNA test at Screening
15. Negative hepatitis C antibody (anti-HCV) test at Screening or positive test followed by a negative HCV RNA test at Screening
16. Able to undergo brain MRI with and without contrast
17. People of childbearing potential must agree to use a highly effective contraceptive method (with a failure rate of < 1%) during study treatment and for at least 6 months following the last dose of study drug and agree not to donate eggs (ova, oocytes) for the purpose of reproduction for the same time period. Acceptable methods of contraception are:

    * Combined estrogen and progestin containing hormonal contraception associated with inhibition of ovulation given orally, intravaginally, or transdermally
    * Progestin-only hormonal contraception associated with inhibition of ovulation given orally, by injection, or by implant
    * Intrauterine device: Intrauterine hormone-releasing system
    * Bilateral tubal occlusion
    * Vasectomised partner
    * Sexual abstinence: Considered a highly effective method only if defined as refraining from heterosexual intercourse during an entire period of risk associated with the study treatment. The reliability of sexual abstinence needs will be evaluated in relation to the duration of the study and to the usual lifestyle of the patient Note: People are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or tubal ligation at least 6 weeks ago. In the case of oophorectomy alone, only when the reproductive status of the person has been confirmed by follow-up hormone level assessment are they considered not of childbearing potential.
18. Sexually active patients that are able to produce a sperm, must use a condom during intercourse and must agree to refrain from sperm donation, from registration on the study until 3 months after the last dose of treatment
19. People of childbearing potential must have a negative highly sensitive serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) at the time of screening and within 48 hours of starting the study drug(s)
20. Ability to adhere to the study visit schedule and all protocol requirements

Exclusion Criteria:

1. Tumors where a gross total resection is not considered feasible by the treating neurosurgeon
2. Tumor involves cerebellum, brainstem, or deep basal ganglia
3. Patients who require urgent resection for mass effect, cerebral edema, or hydrocephalus in the opinion of the treating neurosurgeon
4. Patients with contraindications to MRI or unwilling to undergo MRI
5. History of CNS bleeding as defined by stroke within 6 months prior to registration
6. Contraindication to surgery
7. Treatment with immunosuppressive medications Note: Low-dose corticosteroids (≤ 2 mg/day dexamethasone or equivalent) for tumor-associated edema is permitted. Patients who require corticosteroids > 2mg/day dexamethasone (or equivalent) for acute emergencies during the screening window will be eligible, if the corticosteroid dosing reduces to ≤ 2 mg/day dexamethasone (or equivalent) at least one day prior to the initial trial-mandated biopsy.
8. Active autoimmune disease or immune deficiency including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis
9. Active tuberculosis
10. Patient has had a previous SARS-CoV-2 infection either suspected or confirmed within 4 weeks prior to screening. Acute symptoms must have resolved and based on treating physician's assessment, there are no sequelae that would place the patient at a higher risk of receiving trial treatment
11. Evidence of acute intracranial/intra-tumoral hemorrhage, which requires urgent intervention
12. Severe infection within 4 weeks prior to registration
13. Treatment with a live, attenuated vaccine within 4 weeks prior to registration, or anticipation of need for such a vaccine during study or within 5 months after final dose of nivolumab and relatlimab
14. Patients with prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin or other malignancies with no evidence of disease for 2 years or more
15. Major surgical procedure, other than for diagnosis, within 4 weeks prior to registration
16. History of idiopathic pulmonary fibrosis, organising pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
17. Patient is pregnant or breastfeeding/chestfeeding
18. Prior allogeneic stem cell or solid organ transplantation
19. Known allergy or sensitivity nivolumab, relatlimab, temozolomide or their excipients
20. Patient has any kind of disorder that, in the opinion of the site PI, may compromise the ability of the patient to give written informed consent and/or to comply with all required study procedures
21. Patients with a history of myocarditis
22. Patient has troponin T (TnT) or I (TnI) > 2 × ULN Note: Patients with TnT or TnI levels between > 1 × to 2 × ULN will be eligible if repeat levels within 24 hours are ≤ 1 × ULN. If TnT or TnI levels are between > 1 × to 2 × ULN within 24 hours, the patient must be evaluated by a cardiologist. When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2 × ULN, the patient must be evaluated by a cardiologist. After cardiologist evaluation, the patient may be eligible if the site PI assesses a favorable benefit/risk
23. Left ventricular ejection fraction (LVEF) < 50% by either echocardiogram (ECHO) or multigated acquisition (MUGA) scan within 6 months prior to registration
24. History or evidence of any other clinically significant disorder, condition, or disease (with the exception of those outlined above) that, in the opinion of the site PI would pose a risk to patient safety or interfere with the study evaluation, procedures or completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2029-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the safety of concomitantly administering nivolumab, relatlimab, RT, and TMZ in MGMT methylated patients by monitoring adverse events utilizing CTC Version 5.0 criteria | From date of registration up to 4 weeks
  Proportion of patients with MGMT methylation who experience an unacceptable toxicity during concomitant nivolumab, relatlimab, RT and TMZ by assessing adverse events reported utilizing CTC Version 5.0 criteria
Assess the feasibility of undertaking a peri-operative study of nivolumab with or without relatlimab in patients with ndGBM (Newly diagnosed Glioblastoma) | From date of registration up to 4 weeks
  Proportion of registered patients who undergo biopsy, receive one cycle of randomized neoadjuvant immunotherapy, and undergo surgery during the neoadjuvant phase of the study, OR undergo biopsy that documents the patient to not have GBM.
  Proportion of randomized patients who receive one cycle of randomized neoadjuvant immunotherapy, and undergo surgery.
Establish the biological activity of nivolumab with or without relatlimab in patients with ndGBM by demonstrating the presence of Tumor-infiltrating lymphocytes (TILs) in the resected tumor | From date of registration up to 2 years
  Changes in TILs in formalin-fixed paraffin embedded (FFPE) tumor sections from biopsy to resection during concomitant nivolumab, relatlimab, RT and TMZ

SECONDARY OUTCOMES:
Describe the toxicity of nivolumab with or without relatlimab in patients with ndGBM following biopsy, and prior to surgery | From date of registration up to 2 years
  Proportion of patients who experience Grade 3+ toxicity during neoadjuvant treatment that is attributable to nivolumab and/or relatlimab utilizing CTC Ver 5.0 to assess toxicity
Assess the safety of planned craniotomy and resection after stereotactic biopsy and treatment with nivolumab with or without relatlimab in patients with ndGBM | From date of registration up to 4 weeks
  30-day morbidity post biopsy or post resection
Assess the safety of nivolumab and relatlimab in combination with standard of care chemoradiation in patients with ndGBM. | From date of registration up to 2 years
  Proportion of patients who experience Grade 3+ toxicity during post-surgery treatment that is attributed to nivolumab and/or relatlimab utilizing CTC Ver 5.0 to assess toxicity
Determine the radiological response to nivolumab with or without relatlimab in ndGBM | From date of registration up to 2 years
  Proportion of patients within each arm with a CR or PR per RANO 2.0 criteria
Describe Overall Survival (OS) and Progression Free Survival (PFS) of patients who have been randomized or assigned (as in the Stage 1 safety lead-in) or randomized (Stage 2) to receive neoadjuvant nivolumab administered with or without relatlimab | From date of registration up to 2 years
  Median OS and median PFS
Assess the safety of planned craniotomy and resection after stereotactic biopsy and treatment with nivolumab with or without relatlimab in patients with ndGBM | From date of registration up to 4 weeks
  30-day mortality post biopsy or post resection
Assess the safety of planned craniotomy and resection after stereotactic biopsy and treatment with nivolumab with or without relatlimab in patients with ndGBM | From date of registration up to biopsy or resection
  Number of days delay until biopsy or resection
Assess the safety of planned craniotomy and resection after stereotactic biopsy and treatment with nivolumab with or without relatlimab in patients with ndGBM | From date of registration up to 4 weeks
  Number of subsequent resections

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Long GV, Shklovskaya E, Satgunaseelan L, Mao Y, da Silva IP, Perry KA, Diefenbach RJ, Gide TN, Shivalingam B, Buckland ME, Gonzalez M, Caixeiro N, Vergara IA, Bai X, Rawson RV, Hsiao E, Palendira U, Phan TG, Menzies AM, Carlino MS, Quek C, Grimmond SM, Vissers JHA, Yeo D, Rasko JEJ, Khasraw M, Neyns B, Reardon DA, Ashley DM, Wheeler H, Back M, Scolyer RA, Drummond J, Wilmott JS, Rizos H. Neoadjuvant triplet immune checkpoint blockade in newly diagnosed glioblastoma. Nat Med. 2025 May;31(5):1557-1566. doi: 10.1038/s41591-025-03512-1. Epub 2025 Feb 27. PMID 40016450